CLINICAL TRIAL: NCT05662319
Title: A Phase 3, Single-arm, Multicenter, Multinational, Open-label, One-way Crossover Study to Investigate the Efficacy and Safety of Fitusiran Prophylaxis in Male Participants Aged ≥ 12 Years With Severe Hemophilia A or B With or Without Inhibitory Antibodies to Factor VIII or IX
Brief Title: A Study to Test a Medicine (Fitusiran) Injected Under the Skin for Preventing Bleeding Episodes in Male Adolescent or Adult Participants With Severe Hemophilia
Acronym: ATLAS-NEO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EFC17574; U1111-1275-9584 (Registry Identifier: ICTRP); 2022-500221-33 (Registry Identifier: CTIS)
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — fitusiran

STUDY DESIGN:
Intervention Model Description: One way cross-over
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): In standard of care (SOC) period, participants will receive on-demand or prophylactic treatment with clotting factor concentrates (CFCs) or bypassing agents (BPAs) for 6 months (from Day -168 to Day -1). In fitusiran treatment period, participants will receive subcutaneous fitusiran prophylaxis once every other month (Q2M) or once monthly (QM) for 36 months (from Day 1 to Day 1009). In case of bleeding events participants will receive IV CFCs or BPAs. Participants may receive Antithrombin concentrate (ATIIIC) as rescue medicine.
  .
  Interventions: Drug: Fitusiran; Drug: Clotting factor concentrates (CFC) or bypassing agents (BPA); Drug: Antithrombin concentrate (ATIIIC)

INTERVENTIONS:
Drug: Fitusiran — Pharmaceutical form: Solution for injection Route of administration: Subcutaneous (SC)
Drug: Clotting factor concentrates (CFC) or bypassing agents (BPA) — * Coagulation factor VIII (ATC code: B02BD02)
  * Coagulation factor IX (ATC code: B02BD04)
  * Coagulation factor VIIa (ATC code: B02BD08)
  * Factor VIII inhibitor bypassing activity (ATC code: B02BD03)
  Pharmaceutical form: Solution for infusion Route of administration: Intravenous (IV)
Drug: Antithrombin concentrate (ATIIIC) — Antithrombin III (ATC code: B01AB02) Pharmaceutical form: Solution for infusion Route of administration: Intravenous (IV)

SUMMARY:
This is a multicenter, multinational, open-label, one-way cross-over, Phase 3, single-arm study for treatment of hemophilia.

The purpose of this study is to measure the frequency of treated bleeding episodes with fitusiran in male adult and adolescent (≥12 years old) participants with hemophilia A or B, with or without inhibitory antibodies to factor VIII or IX who have switched from their prior standard of care treatment.

The total study duration will be up to approximately 50 months (200 weeks, 1 study month is equivalent to 4 weeks) and will include:

* A screening period up to approximately 60 days,
* A standard of care (SOC) period of approximately 6 study months (24 weeks),
* A fitusiran treatment period of approximately 36 study months (144 weeks),
* An antithrombin (AT) follow-up period of approximately 6 study months (24 weeks) but may be shorter or longer depending on individual participants AT recovery.

The frequency for telephone visits will be approximately every 2 weeks. For site visits the frequency will be approximately every 8 weeks during the SOC period and approximately every 4 weeks during the fitusiran treatment period. If applicable and if allowed by local regulation, home and/or remote visits may be conducted during the study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe congenital hemophilia A or B (FVIII <1% or FIX level ≤2%) as evidenced by a central laboratory measurement at screening or documented medical record evidence.
* For participants currently not on prophylaxis (CFC or BPA on-demand): A minimum of 4 bleeding episodes requiring BPA (inhibitor participants) or CFC (non-inhibitor participants) treatment within the last 6 months prior to screening.
* Willing and able to comply with the study requirements and to provide written informed consent and assent in the case of participants under the age of legal consent, per local and national requirements

Exclusion Criteria:

* Known co-existing bleeding disorders other than congenital hemophilia A or B
* History of arterial or venous thromboembolism, not associated with an indwelling venous access
* History of intolerance to SC injection(s).
* Current participation in immune tolerance induction therapy (ITI)
* Prior gene therapy
* Current or prior participation in a fitusiran trial
* Current or prior participation in a gene therapy trial
* Received an investigational drug or device within 30 days prior to the screening visit or within 5 half-lives of the investigational drug (or device) prior to the screening visit, whichever is longer
* Presence of clinically significant liver disease AT activity <60% at Screening
* Co-existing thrombophilic disorder
* Hepatitis C virus antibody positive, except participants who have negative Hepatitis C viral load and no evidence of cirrhosis
* Presence of acute hepatitis, ie, hepatitis A, hepatitis E.
* Presence of acute or chronic hepatitis B infection
* Known to be HIV positive with CD4 count <200 cells/μL.
* Reduced renal function The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2029-01-25 (Estimated)

PRIMARY OUTCOMES:
Annualized bleeding rate (ABR) in the fitusiran primary efficacy period | Day 169 to Day 505 (since the first dose of fitusiran)
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs, e.g., hemarthrosis, muscle, or mucosal bleeding.

SECONDARY OUTCOMES:
Annualized bleeding rate (ABR) while on fitusiran prophylaxis in the fitusiran primary efficacy period and ABR while on prophylaxis standard of care (SOC) in the SOC period | Day 169 to Day 505 (primary efficacy period) and Day -168 to Day -1 (SOC period)
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs, e.g., hemarthrosis, muscle, or mucosal bleeding.
Annualized bleeding rate (ABR) while on fitusiran prophylaxis in the fitusiran primary efficacy period and ABR while on on-demand standard of care (SOC) in the SOC period | Day 169 to Day 505 (primary efficacy period) and Day -168 to Day -1 (SOC period)
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs, e.g., hemarthrosis, muscle, or mucosal bleeding.
Annualized spontaneous bleeding rate in the fitusiran primary efficacy period and in the SOC period | Day 169 to Day 505 (primary efficacy period) and Day -168 to Day -1 (SOC period)
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs, e.g., hemarthrosis, muscle, or mucosal bleeding.
  A spontaneous bleeding episode is a bleeding event that occurs for no apparent or known reason, particularly into the joints, muscles, and soft tissues.
Annualized joint bleeding rate in the fitusiran primary efficacy period and in the SOC period | Day 169 to Day 505 (primary efficacy period) and Day -168 to Day -1 (SOC period)
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs, e.g., hemarthrosis, muscle, or mucosal bleeding.
  A joint bleeding episode is characterized by an unusual sensation in the joint ("aura") in combination with 1) increasing swelling or warmth over the skin over the joint, 2) increasing pain, or 3) progressive loss of range of motion or difficulty in using the limb as compared with baseline.
Change in Haem-A-QOL physical health score and total score during SOC and during fitusiran prophylaxis | Day 1 (D1) to Day 505, and from D1 to Day 1009, and during SOC from Day-168 to D-1
  The Haem-A-QoL will be provided to participants ≥17 years of age and includes 46 items contributing to 10 QoL domains (physical health, feelings, view of yourself, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, partnership, and sexuality). Scoring for each item is based on a 5-point Likert scale (never, rarely, sometimes, often, and all the time), and higher scores represent greater impairment.
Annualized bleeding rate (ABR) in the fitusiran 18-month efficacy period | Day 1 to Day 505
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs, e.g., hemarthrosis, muscle, or mucosal bleeding.
Annualized bleeding rate (ABR) in the fitusiran 36-month treatment period | Day 1 to Day 1009
  A bleeding episode is defined as any occurrence of hemorrhage that requires administration of CFCs or BPAs, e.g., hemarthrosis, muscle, or mucosal bleeding.
Annualized weight-adjusted consumption of CFC/BPA | Day -168 until Day 1009
  All CFC or BPA doses (including doses per kg body weight) administered during the study treatment will be recorded
Number of participants with adverse events | Date of signed ICF (Day -228 to Day -169) until last visit (approximately 50 months after date of signed ICF)
  All AEs (serious or nonserious) will be collected from the signing of the informed consent form (ICF) until last AT follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (50):
- United States (8):
  - Center for Inherited Blood Disorders (CIBD) Site Number : 8400012, Orange, California
  - M Health Fairview University of Minnesota Medical Center - West Bank- Site Number : 8400016, Minneapolis, Minnesota
  - Hackensack University Site Number : 8400009, Hackensack, New Jersey
  - Northwell Health Hemostasis and Thrombosis Center Site Number : 8400015, New Hyde Park, New York
  - University Hospitals of Cleveland Site Number : 8400001, Cleveland, Ohio
  - UPMC Children's Hospital of Pittsburgh-4401 Penn Ave Site Number : 8400017, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas- Site Number : 8400018, Dallas, Texas
  - Gulf States Hemophilia and Thrombophilia Center- Site Number : 8400002, Houston, Texas
- Canada (3):
  - Investigational Site Number : 1240001, Hamilton, Ontario
  - Investigational Site Number : 1240002, Hamilton, Ontario
  - Investigational Site Number : 1240004, Toronto, Ontario
- China (3):
  - Investigational Site Number : 1560003, Beijing
  - Investigational Site Number : 1560001, Guangzhou
  - Investigational Site Number : 1560002, Jinan
- France (3):
  - Investigational Site Number : 2500003, Le Kremlin-Bicêtre
  - Investigational Site Number : 2500002, Lille
  - Investigational Site Number : 2500001, Paris
- Germany (2):
  - Investigational Site Number : 2760001, Berlin
  - Investigational Site Number : 2760002, Hamburg
- Greece (2):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000002, Athens
- India (5):
  - Investigational Site Number : 3560004, Bangalore
  - Investigational Site Number : 3560007, Bhubaneswar
  - Investigational Site Number : 3560001, Pune-411011
  - Investigational Site Number : 3560006, Punjab
  - Investigational Site Number : 3560003, Vellore
- Italy (2):
  - Investigational Site Number : 3800003, Rozzano, Milano
  - Investigational Site Number : 3800001, Milan
- Japan (3):
  - Investigational Site Number : 3920003, Nagoya, Aichi-ken
  - Investigational Site Number : 3920001, Kashihara-shi, Nara
  - Investigational Site Number : 3920002, Saitama-shi, Saitama
- Mexico (3):
  - Investigational Site Number : 4840002, Monterrey, Nuevo León
  - Investigational Site Number : 4840004, Chihuahua City
  - Investigational Site Number : 4840001, Veracruz
- Poland (3):
  - Investigational Site Number : 6160002, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160004, Lodz, Lódzkie
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
- Investigational Site Number : 6820002, Jeddah, Saudi Arabia
- South Africa (2):
  - Investigational Site Number : 7100003, Johannesburg
  - Investigational Site Number : 7100001, Parktown
- South Korea (2):
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (2):
  - Investigational Site Number : 7240002, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number : 7240003, Zaragoza
- Taiwan (2):
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580003, Taipei
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920002, Adana
  - Investigational Site Number : 7920004, Akdeniz
  - Investigational Site Number : 7920001, Çapa
  - Investigational Site Number : 7920003, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17574 Plain Language Results Summaries — https://www.trialsummaries.com/Study/StudyDetails?id=25264&tenant=MT_SNY_9011